CLINICAL TRIAL: NCT01327677
Title: Post Craniotomy Analgesia Safety Monitoring With ET CO2
Brief Title: Safety Study of Analgesia After Craniotomy Surgery With End Tidal (ET) Carbon Dioxide (CO2) Monitoring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00029336
Record Dates: First submitted 2011-03-25; First posted 2011-04-01 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: pain management; opioid analgesic therapy; safety; craniotomy
MeSH Terms: conditions — Pain; Agnosia | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pro re nata (PRN) fentanyl (Active Comparator): A nurse can give the patient up to 3 doses of fentanyl intravenously (through a vein) each hour whenever a patient indicates that he or she is in pain.
  Interventions: Drug: Fentanyl
- Intravenous Patient-controlled Analgesia (IVPCA) fentanyl (Active Comparator): Fentanyl will be given with a Patient Controlled Analgesia (PCA) pump.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — 25-50 mcg every 20 minutes
  Other Names: Fentanyl PRN
  Arms: Pro re nata (PRN) fentanyl
Drug: Fentanyl — 20mcg/demand dose with an 8 minute lock out
  Other Names: Fentanyl PCA
  Arms: Intravenous Patient-controlled Analgesia (IVPCA) fentanyl

SUMMARY:
This research is being done to compare two methods of giving fentanyl, a narcotic often given to patients following brain surgery and determine if one method has more side effects than the other. Both of these methods are available in the postoperative treatment of pain. This research also is being done to determine if patients receiving narcotic pain medicine will benefit from additional monitoring of carbon dioxide levels. Since narcotic pain medicines can slow down breathing, The investigators want to see if measuring exhaled carbon dioxide levels will help identify a slower breathing rate and improve safety.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female, English speaking patients undergoing supratentorial craniotomy for tumor under general anesthesia at the Johns Hopkins Hospital will be eligible for this study.

Exclusion Criteria:

* pregnant women
* patients with post operative neurological changes
* patients who remain intubated post-operatively
* patients who require the use of concomitant administration of sedatives

  * patients who are unable to initiate a PCA bolus
  * patients who are unable to communicate verbally
  * patients who are allergic to fentanyl
* patients who have a history of narcotic abuse
* patients who have a history of chronic pain requiring opioids
* patients who have been in any investigational drug trial within 1 month of the treatment day
* patients who have chronic respiratory insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athir H Morad, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PRN Fentanyl: A nurse can administer up to 3 doses of fentanyl intravenously (through a vein) each hour whenever a patient indicates that he or she is in pain.
  Fentanyl: 25-50 mcg every 20 minutes
- PCA Fentanyl: A patient can self-administer fentanyl intravenously using a Patient Controlled Analgesia (PCA) pump.
  Fentanyl: 20mcg/demand dose with an 8 minute lock out
Period: Overall Study
Arm/Group | PRN Fentanyl | PCA Fentanyl
Started | 68 | 69
Completed | 48 | 56
Not Completed | 20 | 13

BASELINE CHARACTERISTICS:
Groups:
- IVPCA Fentanyl: A patient can self-administer fentanyl intravenously with a Patient Controlled Analgesia (PCA) pump.
  Fentanyl: 20mcg/demand dose with an 8 minute lock out
- Total: Total of all reporting groups
Arm/Group | PRN Fentanyl | IVPCA Fentanyl | Total
Number analyzed (Participants) | 48 | 56 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: As the result of patients either not completing the assigned intervention due to premature withdrawal from the protocol, protocol violations, or incomplete data capture, the number of analyzed patients was reduced compared to the originally allocated number.
  years | 49.1 (14.0) | 50.4 (13.7) | 49.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: As the result of patients either not completing the assigned intervention due to premature withdrawal from the protocol, protocol violations, or incomplete data capture, the number of analyzed patients was reduced compared to the originally allocated number.
  Participants
    Female | 26 | 25 | 51
    Male | 22 | 31 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: As the result of patients either not completing the assigned intervention due to premature withdrawal from the protocol, protocol violations, or incomplete data capture, the number of analyzed patients was reduced compared to the originally allocated number.
  Participants
    White | 42 | 44 | 86
    Black | 5 | 7 | 12
    Other | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Depression
Description: Defined by minimum respiratory rate (breaths/minute).
Time Frame: up to 24 hours postoperatively
Measure: Mean (Standard Error); unit: breaths/minute
Groups:
- PCA Fentanyl: A patient can self-administer fentanyl intravenously with a Patient Controlled Analgesia (PCA) pump.
  Fentanyl: 20mcg/demand dose with an 8 minute lock out
Arm/Group | PRN Fentanyl | PCA Fentanyl
Number analyzed (Participants) | 48 | 56
breaths/minute | 10.9 (0.4) | 10.5 (0.4)

2. Primary Outcome: Respiratory Depression
Description: Defined by maximal End Tidal CO2 (mmHg)
Time Frame: Up to 24 hours postoperatively.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- (Pro re Nata) PRN Fentanyl: A nurse can give the patient up to 3 doses of fentanyl intravenously (through a vein) each hour whenever a patient indicates that he or she is in pain.
  Fentanyl: 25-50 mcg every 20 minutes
Arm/Group | (Pro re Nata) PRN Fentanyl | Intravenous Patient-controlled Analgesia (IVPCA) Fentanyl
Number analyzed (Participants) | 48 | 56
mmHg | 41.4 (0.6) | 41.1 (0.7)

3. Secondary Outcome: Hypoxia
Description: Defined by minimum oxygen saturation (SaO2)
Time Frame: up to 24 hours postoperatively
Measure: Mean (Standard Error); unit: Percent Oxygen Saturation
Arm/Group | PRN Fentanyl | PCA Fentanyl
Number analyzed (Participants) | 48 | 56
Percent Oxygen Saturation | 95.8 (0.2) | 96.3 (0.2)

4. Other Pre Specified Outcome: Mean Fentanyl Consumption
Description: Amount of cumulative fentanyl consumed in mcg
Time Frame: up to 24 hours postoperatively
Measure: Mean (Standard Error); unit: micrograms/ hour
Arm/Group | PRN Fentanyl | PCA Fentanyl
Number analyzed (Participants) | 48 | 56
micrograms/ hour | 16.5 (2.65) | 26.4 (2.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of patient enrollment in the Neurosciences Critical Care Unit, within 24 hours of surgery.
Arm/Group | PRN Fentanyl | PCA Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/56
Other Adverse Events (participants affected / at risk) | 0/48 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes